CLINICAL TRIAL: NCT02673450
Title: PER3 Clock Gene Polymorphism, Clock Gene Expression and Delirium in the Intensive Care Unit. A Prospective Cohort Study.
Brief Title: PER3 Clock Gene Polymorphism, Clock Gene Expression and Delirium in the Intensive Care Unit.
Status: Withdrawn | Type: Observational
Why Stopped: Lack of lab ressources
Sponsor: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Stine Estrup, Ph.d. student MD, Zealand University Hospital
Other Study IDs: SE 2-16
Record Dates: First submitted 2016-02-01; First posted 2016-02-04 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 21 ml of blood from each patient is kept in a biobank for 10 years
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study investigates a possible relationship between disturbance of the cyclic expression of ten different clock genes and development of delirium in patients admitted to an intensive care unit

It also investigates a possible relationship between disturbance of the cyclic expression of melatonin and development of delirium in patients admitted to an intensive care unit.

Finally a possible relationship between genetic differences in the PER3 gene and development of delirium is investigated.

DETAILED DESCRIPTION:
An increasing number of patients are treated at ICUs worldwide. The majority of these patients survive critical illness and are discharged from hospital. In recent decades, improved therapy and survival at ICUs has increased focus on long term outcomes and post-ICU rehabilitation. Both physical and mental problems following admission for ICU therapy can be found for years after discharge. It is therefore important to discover factors that may have a significant impact for a worsened outcome, in order to prevent and treat these impairments.

Cognitive deficiencies may affect large proportions of the post intensive care population and mild cognitive impairment was demonstrated for up to 40% of the patients when evaluated three months after discharge. Recovery was slow and at one year follow up, 25% of the patients still showed impairment comparable to mild traumatic brain injury.

The presence of delirium during ICU stay has been associated with a worsened cognitive outcome at both 3 and 12 months follow up. Both patient's global cognition and especially executive function was impaired. Furthermore, a longer duration of the delirium period was associated with a poorer cognitive function. Incidence of delirium has also shown association to higher mortality rates and a longer hospital stay when compared to patients without delirium. In previous studies, the second day of admission has had the highest incidence of delirium.

Alterations in sleep architecture with a more shallow sleep and disruptions of the sleep wake cycle, is common in both ICU patients and patients with delirium. Sleep deprivation is often seen in delirious patients, and consequently, it has been suggested to be a risk factor for development of delirium.

The circadian rhythm is an inborn cycle of biological activity based on 24 hour intervals, and the rhythmicity interacts with sleep homeostasis in order to regulate sleep-wake cycles of individuals. In humans, the circadian rhythm is controlled by the suprachiasmatic nucleus (SCN) (the circadian clock) mediating melatonin secretion from the pineal gland to regulate the sleep-wake cycle. A number of factors, especially daylight, influence the SCN.

When blue light (460-480 nm wavelengths) reaches the retina and excites photoreceptors, it communicates with the pineal gland and secretion of melatonin is reduced to a minimum. Melatonin is secreted at night when blue light is absent and promotes sleep by activation of melatonin receptors. Melatonin secretion also interacts with a number of body functions, including core body temperature and the cardiac and immune systems. It is one of the key molecules in circadian rhythmicity. The circadian rhythm is not only affected by light, but is also synchronized by other factors, including shift work, artificial light exposure and exercise.

A number of genetic markers known as clock genes play a major role in the circadian control of different processes in the body. These genes may determine an individual's chronotype (morningness/eveningness), sensitivity to sleep disturbance and sleep deprivation, but much of their significance and function is still unknown.

A group of genes named PERIOD genes are shown to be involved in determining individual sleep wake regulation. PERIOD3 (PER3) is found in three subtypes: PER3 4/4, PER3 4/5 and PER3 5/5. The numbers refer to a variable number of tandem repeat polymorphism where a motif of 54 nucleotides is repeated for 4 or 5 U. Studies in large populations have shown 10% of individuals to be homozygous for the 5'-variation, 50% for the 4'-variation and 40% to be heterozygous.

Patients with homozygosity of the long allele (PER35/5) have more slow wave sleep and longer sleep duration compared to the other sub-types. Though no difference in melatonin or cortisol levels where seen, the two types reacted very differently to sleep deprivation. PER35/5 individuals performed poorly on a variety of cognitive tests compared to PER34/4. This information might help to identify subgroups of patients especially sensitive to development of delirium.

A recent study explored the relationship between PER3 genotype and postoperative cognitive dysfunction and did not find an association. The distribution of PER3 subtypes were as expected from previous studies. However, a possible association between PER 3 genotypes and cognitive dysfunction has never been investigated in ICU patients.

A number of other genes are involved in the circadian rhythm. These genes are expressed in a rhythmic manner following the natural light/dark cycle.

In healthy subjects, severely disturbed expression of the clock genes Clock, Cry1-2, Per1-3, Rorα, Bmal1, Rev-erb and CSNK1ε has been demonstrated after injection of endotoxin.

In septic ICU patients, a desynchronised expression of Cry-1 and Per-2 has been demonstrated. This disturbance was linked to secretion of proinflammatory cytokines as tumor necrosis factor α (TNFα) and interleukin 6 (IL-6).

The implication of the above is that if a disturbed circadian rhythm can be demonstrated to be associated with patients in delirium, we might in the future be able to identify patients with a higher risk of developing delirium - even in comatose or heavily sedated patients. Something which is not possible with the current diagnostic methods.

In this study, we therefore wish to investigate the relationship between PER3 gene polymorphism and incidence of delirium. This may help to identify patient groups at a higher risk of developing delirium and potentially prevent or treat these patients at an earlier stage.

The other objective is to identify differences in melatonin and cyclic gene expression in delirious patients, compared to other critically ill patients. This may be a new perspective for the diagnosis of delirium in heavily sedated patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age admitted to the ICU at Køge Hospital in the study period

Exclusion Criteria:

* Not able to speak or understand Danish
* Melatonin (ATC N05CH01) or melatonin agonist (ATC N06AX) treatment prior to admission
* Known insomnia (daily hypnotic (ATC N05C) consumption or known sleep disorder)
* Patients discharged from the ICU during the test period (time from first to last blood sample)
* Patients who die during the test period
* Patients transferred to another hospital during ICU stay

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the ICU at Køge Hospital in the study period
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Clock gene expression | 24 hours
  Association between expression of clock genes (Clock, Cry1-2, Per1-3, Rorα, Bmal1, Rev-erb and CSNK1ε) (measured at 6am, 10am, 2pm, 6pm, 10pm and 2am) and incidence of delirium at the ICU

SECONDARY OUTCOMES:
Melatonin secretion | 24 hours
  Association between secretion of melatonin at 6am, 10am, 2pm, 6pm, 10pm and 2am. Cosinor curve analysis (mesor, amplitude and acrophase) and incidence of delirium
PER3 subtype | 24 hours
  Association between PER3 subtype determination at 6am (PER3 4/4, PER3 4/5 and PER3 5/5) and incidence and duration of delirium
Delirium type | 24 hours
  Delirium type (hypoactive/hyperactive/mixed) associated to PER3 and expression pattern of clock genes and melatonin secretion
Demographic variables | 24 hours
  Age, gender, weight at admission associated to PER3 and expression pattern of clock genes and melatonin secretion
Sedation | 24 hours
  Infusion of propofol, dexmedetomidine, midazolam, sufentanil, remifentanil associated to PER3 and expression pattern of clock genes and melatonin secretion
Disease severity | 24 hours
  SAPS II score at admission associated to PER3 and expression pattern of clock genes and melatonin secretion
Admission type | 24 hours
  Type of admission (medical/acute surgical/elective surgical) associated to PER3 and expression pattern of clock genes and melatonin secretion
Length of stay | Up to 6 months
  Length of stay at ICU and hospital associated to PER3 and expression pattern of clock genes and melatonin secretion
Number of ventilator days | Up to 6 months
  Number of ventilator days at ICU and hospital associated to PER3 and expression pattern of clock genes and melatonin secretion
ICU delirium | Up to 6 months
  Delirium defined as positive CAM-ICU or treatment with antipsychotics

CONTACTS AND LOCATIONS:
Overall Officials: Ole Mathiesen, MD, PhD, Study Chair — Køge Hospital
Locations (1):
- Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No